CLINICAL TRIAL: NCT03445052
Title: The XPAND Evaluation of a Personalised Adherence Intervention to Improve Photoprotection Behaviour in Adults With Xeroderma Pigmentosum (XP): Randomised Controlled Trial.
Brief Title: XPAND Trial: Enhancing XP Photoprotection Activities - New Directions
Acronym: XPAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Newcastle University (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 236877
Record Dates: First submitted 2018-02-07; First posted 2018-02-26 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Xeroderma Pigmentosum
Keywords: Adherence; Behaviour change; Intervention; Photoprotection; Ultraviolet radiation
MeSH Terms: conditions — Xeroderma Pigmentosum

STUDY DESIGN:
Intervention Model Description: The study will test the efficacy of the intervention using a randomised controlled trial design. It is a "delayed RCT", one group will receive the intervention in year 1 and be compared to the other "control group" in year 2. The control group will receive the intervention in year 2. The UVR dose to the face will be measured at baseline (21 days in March -April 2018) and will then be assessed at two follow-up periods in 2018 (June to July; August to September); two periods in 2019 (delayed intervention group). Psychosocial constructs will be measured by self report questionnaires at baseline and at the start of each UVR measurement period, as well as daily during these episodes. 9 months after baseline self-report questionnaires will be completed. A qualitative process evaluation will be conducted after the intervention is complete. A health economic evaluation of the intervention will be assessed by completion of HRQOL and service use questionnaires in December 2018, 2019.
Who Masked: Outcomes Assessor
Masking Description: Group Allocation will be concealed from the statisticians conducting the analysis until the analysis relevant to the primary study objective has been completed.
  Care providers: Group allocation will be concealed from the XP clinical team who are not part of the research team. This is to avoid change in the standard care of these participants during the trial (i.e., greater/less discussion of adherence to photoprotection during the routine clinical appointment). Randomisation will be broken if the intervention facilitator is concerned about the participant's emotional wellbeing at any point during delivering the intervention. In this case the clinical team will be alerted and the participant will be referred to the clinical psychologist at the XP service for assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2018 XPAND Intervention Arm (Experimental): This group will receive the personalised adherence intervention in 2018 in addition to routine clinical care.
  Interventions: Behavioral: XPAND
- 2018 XPAND Control Arm (No Intervention): This group will receive routine clinical care and act as the control group for the primary objective: To compare the mean daily dose of UVR (SEDs) reaching the face between the intervention group and control group over a 3 week period in June to July (follow-up 1). This group will receive the intervention in 2019, to allow within group change to be assessed.

INTERVENTIONS:
Behavioral: XPAND — The intervention is personalised to the psychosocial factors influencing poor photoprotection for each person. These factors could include beliefs that reduce motivation to protect as well as factors that prevent intentions being translated into action. The facilitator will use behaviour change techniques to target the factor most important for each person. Standardised content related to habit formation will be received. The intervention will be delivered via 7 1:1 sessions with a facilitator (psychologists or clinical nurse specialist). Sessions 1 (1.5 hours maximum) and 6 (45 minutes) will be delivered face to face in the home of the participant and the remaining sessions will be conducted via telephone calls or skype sessions.
  Arms: 2018 XPAND Intervention Arm

SUMMARY:
People with Xeroderma Pigmentosum (XP) have a genetic condition which stops their skin repairing damage from Ultraviolet Radiation (UVR). This means they are much more likely to develop potentially fatal skin cancers. The only way to reduce this damage is to rigorously protect the skin, by limiting UVR exposure. This done in a number of ways including: staying indoors; wearing protective clothing, sunscreen and glasses. People with XP can find it difficult to maintain this level of protection, putting themselves at risk.

This research will test whether an intervention designed to enhance photoprotection activities is successful. It will use a randomised controlled trial design to compare the amount of UVR reaching the face, between participants receiving the intervention and those receiving standard clinical care. The amount of UVR reaching the face is important, as this is where people with XP develop most cancers. It is dependent on the overall level of exposure to UVR in the environment, and photoprotection used.

The intervention involves a tailored conversation with the participant about their photoprotection practices. It will target both the overall exposure to UVR and the photoprotection used when outdoors, and will be conducted in 7 sessions with an intervention facilitator. The content will be dependent on the specific photoprotection behaviour being targeted (e.g., poor sunscreen application) and the reasons for poor photoprotection for each person. This could be low motivation related to doubts about the need to protect and concerns about protecting. Other barriers to protection might be lack of routines. The facilitator will provide information tailored to these beliefs and use other standard behaviour change techniques to encourage the development of "better" photoprotection habits.

The investigators predict that the intervention group will have a lower mean daily dose of UVR to the face compared to the control group in two time periods in the summer months.

DETAILED DESCRIPTION:
Xeroderma Pigmentosum (XP) is a rare autosomal recessive inherited condition caused by defective Nucleotide Excision Repair. Patients may develop skin cancers from childhood onwards, ocular damage, and neurological deterioration. The clinical management of XP relies on minimising exposure of the skin to Ultraviolet radiation (UVR), which is the only means of preventing skin cancer and eye disease. Reduction in UVR exposure is achieved by a combination of lowering overall exposure and rigorously photoprotecting when outdoors. This involves wearing protective clothing and application of factor 50 sunscreen to any exposed skin. Evidence from new research carried out by our team, indicated that photoprotection was inadequate with room for improvement. The clinical consequence of this sub-optimal photoprotection is higher incidence of skin cancers, including malignant melanoma, which require surgery and can be life threatening.

The investigators have designed a personalised adherence intervention, using a systematic approach called Intervention Mapping, to target the determinants of UVR reaching the face. The intervention will not require advanced therapeutic skills and has been designed to be delivered by a range of healthcare professionals. It will be tailored to the predictors of photoprotection, relevant for each person, and will be delivered via seven one-to-one sessions between the intervention facilitator and patient. Sessions 1 and 6 will be delivered face to face in the home and the remaining sessions will be conducted via telephone calls or skype sessions, depending on the preference of the participant. The facilitator will use a range of behaviour change techniques to target each determinant relevant to each individual, alongside generic components to promote habit and planning which will be delivered to all. Personalised text messages, sunscreen application video and activity sheets will also be used. The intervention facilitator will use the collaborative conversational style of Motivational Interviewing.

The primary objective is to test the efficacy of a personalised adherence intervention to reduce the level of UVR reaching the face by improving adherence to UVR protection advice.

Primary objective

1. To compare the mean daily dose of UVR (SEDs) reaching the face between the intervention group and control group over a 3 week period in June to July (follow-up 1) Secondary objectives

1. To compare the mean daily dose of UVR (SEDs) reaching the face between the intervention group and control group in August to September 2018 (follow-up 2)
2. To compare photoprotection practices between the intervention group and control group in June to July (follow-up 1)
3. To compare photoprotection practices between the intervention group and control group in August to September (follow-up 2)
4. To investigate with-in group changes in photoprotection practices pre and post the intervention up to 9 months follow-up
5. To compare between group differences in mean mood, habit formation, goal priority and self-efficacy for managing barriers between the intervention group and control group in June to July (follow-up 1)
6. To compare between group differences in mean mood, habit formation, goal priority and self-efficacy for managing barriers between the intervention group and control group in August to September (follow-up 2)
7. To investigate with-in group changes in quality of life, emotional wellbeing, habitual behaviour, self-efficacy, personalised psychosocial drivers, self-rated adherence pre and post the intervention up to 9 months follow-up
8. To qualitatively explore psychosocial "mechanisms of change" related to the intervention from the perspective of the participant
9. To qualitatively explore the acceptability and feasibility of the intervention from the perspective of the participant
10. To identify the health economic cost of the intervention

Design The study will test the efficacy of the intervention using a randomised controlled trial (RCT) design. It is a "delayed RCT", the intervention group will receive the intervention in year 1 (2018) and be compared to the control group. The control group will receive the intervention in 2019. It would not be possible to complete the intervention and measurement in both groups during the same season, when UVR levels are comparable. The UVR dose to the face will be measured at baseline (21 days in March -April 2018) and will then be assessed at two follow-up periods of 21 days in 2018 (June to July; August to September) and two follow-up periods in 2019 (March, June to July) (delayed intervention group only). Psychosocial constructs and photoprotection practices will be assessed at baseline, at the start of each follow-up period (self-report questionnaires) and during these follow-up periods (daily measures on the UVR protection diary). 9 months after baseline (December 2018, 2019) self-report questionnaires will be completed. A process and acceptability evaluation will be conducted using qualitative interviews. A health economic evaluation of the intervention will be assessed by completion of questionnaires to assess health-related quality of life and service use in December 2018, 2019. The study is a main trial. There is no pilot or feasibility study due to the small population from which the sample will be obtained (adults with XP in UK without cognitive impairment).

Procedure Eligible patients will be identified from the patient list, XP Service at Guy's and St Thomas' NHS Foundation Trust and sent an invitation letter. The investigators will send out the information sheet and request that the patient contact the research team if they wish to participate. This will be followed up with a phone call answer any questions they might have and see if they wish to participate. Those wishing to take part will be visited by a member of the research team to complete the consent process and deliver study materials. Participants will complete the baseline assessment which involves wearing a UVR monitor called a dosimeter, completing a UVR protection diary for a 3 week period (March-April 2018) and questionnaires. The dosimeter is then worn continuously during the day March to September 2018. Participants are then randomised to receive the intervention in 2018 or 2019. Participants receiving the intervention in 2018, will then take part in the first 6 sessions of the intervention across 12 weeks. All participants then repeat the baseline measurement protocol. The intervention group will then receive a booster intervention session and both groups will complete a second follow-up assessment period. Intervention participants will then take part in a qualitative interview. At 9-months post baseline all participants will complete self-report questionnaires. If a participant is randomised to receive the intervention in 2019, they will repeat the procedure excluding the second follow-up assessment period and will wear the dosimeter from March to July 2019.

Data management To protect the anonymity of the participants, once consent has been given, participants will be given a unique identifier. Data recorded on paper will be stored at the XP research office at King's College London., in locked cabinets in a locked room. Data entered electronically will be stored in password protected files accessible via a drive only accessible to the XP Research Team.

Progress will be monitored by the Trial Steering Committee, Independent Steering Committee and our funder NIHR.

Sample size The target sample size is 24 accounting for potential attrition of 20%. Based on the primary outcome being the between group difference in mean daily UVR dose to the face across a period of 21 days in June to July, the target sample size of 20 individuals (excluding dropouts) leads to a total of 210 daily observations for the 10 participants randomised to each arm. In previous research, the mean daily UVR dose to the face was .27 SED (SD=.14) with a within-person correlation of ICC=.31. Adjusting for the design effect due to the dependence of assessments within individuals, and accepting a liberal 10% alpha and 20% beta level due to the rare nature of the condition, this sample size would have 80% power to detect a reduction of .10 SED in mean UVR dose to the face. In terms of standardised mean difference this relates to an effect size of d=.73, which is considered to be a large effect. Given the tailored nature and expected intensity of the intervention, expecting such a difference does not seem unreasonable though it must be accepted that power would not be sufficient to detect smaller but still clinically meaningful differences. Where the target dose to the face is 0 SED, a reduction of .1 SED relates to around a 30% overall reduction in UVR dose to the face. To allow for an estimated attrition rate of 20% the target total sample size is 24.

Analysis for primary objective The treatment effect on the primary outcome of daily UVR dose to the face during over 21 days between June and July and secondary outcome of daily UVR dose to the face during over 21 days between August and September will be estimated using generalised linear mixed models. Given the skewed distribution of UVR dose to face a logarithmic transformation will be applied. A random intercept will account for the repeated assessments of UVR dose to the face within individuals across 42 days. Group will be entered as an indicator variable along with a time period indicator (i.e. early vs late summer), any stratification factors used in the randomisation (e.g. complementation type) and baseline mean daily UVR dose to face. Two baseline levels of mean daily UVR dose to face will be included in the analysis as covariates; mean daily UVR dose to face collected in previous study (21 days between June and July 2016) and pre-intervention mean daily UVR dose to face ( 21 days between March and April 2018). Given the rare nature of the condition, the investigators will accept a higher than usual false positive rate and will accept the treatment is efficacious where the p-value for the group coefficient is p<.1 (i.e. 10% critical alpha level). The analysis will follow the intention to treat principle with individuals analysed within the groups to which they were randomised irrespective of whether they received or persisted with the intervention. Sensitivity analysis will consider treatment effects in a per-protocol analysis of those completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis (on the basis of DNA repair study results) of Xeroderma Pigmentosum
2. Age >16 years
3. Sub-optimal adherence to photoprotection when outdoors, identified by clinical team from data held in medical notes.

For those who participated in our previous research study, sub-optimal adherence will be confirmed from data collected during that study. They will be eligible if they meet any of the following criteria:

1. Score <20 on the Adherence to Photoprotection scale (total score is 25 - optimal protection) from a cross-sectional questionnaire completed during our previous research.
2. Using photoprotective clothing that have been assessed by the clinical team as anything other than "very good or excellent" on anytime outdoors, recorded on the daily UVR protection diary.
3. Having a "resistant" mode of adjustment to photoprotection in the qualitative analysis

Exclusion Criteria:

1. Adults diagnosed with cognitive impairment
2. Adults with inadequate English to be able to converse with the intervention facilitators
3. Adults diagnosed with current clinical depression or anxiety

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Mean daily dose of ultraviolet radiation (UVR) to the face using a dosimeter and diary. | It will measured in all participants for 21 days at 10 weeks post baseline
  The mean daily dose of UVR will be calculated by combining data from: (i) A UVR recorder wrist-worn device, (dosimeter) (ii) Patients' photoprotective activities self-monitored and recorded on a diary. The dosimeter provides real-time measurements of ambient UVR. It measures UVR in units of Standard Erythemal Dose (SEDs), every 5 seconds and records the mean every 5 minutes. The diary has a grid format with the day split into 15 minute segments. Participants record time spent outside rounded to the nearest 15 minutes and their photoprotection activity (e.g. hat, hoodie worn-up) during that time. During each 15 minute interval the dose of UVR to the face (in SEDs) equals the UVR exposure recorded by the dosimeter weighted by the protection associated with photoprotection behaviours recorded for that interval on the diary. Weights will be generated based on the degree of photoprotection afforded by each activity.

SECONDARY OUTCOMES:
Mean daily mood | It will measured in all participants for 21 days at 3 time periods: baseline, 10 weeks and 16 weeks post baseline. The control group will complete a 21 day follow-up at 12 months (52 weeks) and 14.5 months (62 weeks) post baseline.
  This is a self reported measure of mood. It will be measured daily by completion of a single question designed for the study. The question is: How would you describe your mood today? (0= very negative - 10=very positive). Participants respond by marking a number between 0 and 10. A higher score indicates a more positive mood. Mean daily mood will be recorded across each 21 day measurement period for each participant.
Mean daily automaticity of UVR protection activity | It will measured in all participants for 21 days at 3 time periods: baseline, 10 weeks and 16 weeks post baseline. The control group will complete a 21 day follow-up at 12 months (52 weeks) and 14.5 months (62 weeks) post baseline.
  This is a self reported measure of automaticity. It will be measured daily by completion of a single question designed for the study, adapted from the Self-Report Behavioural Automaticity Index (SRBAI). The question is: How much do you agree that UVR protection of your face today was something you did automatically without thinking? (0=strongly disagree - 10= strongly agree) Participants respond by marking a number between 0 and 10. A higher score indicates greater automaticity. Mean daily automaticity will be recorded across each 21 day measurement period for each participant.
Mean daily prioritisation of UVR protection activity | It will measured in all participants for 21 days at 3 time periods: baseline, 10 weeks and 16 weeks post baseline. The control group will complete a 21 day follow-up at 12 months (52 weeks) and 14.5 months (62 weeks) post baseline.
  This is a self reported measure of prioritisation of UVR protection activity compared to other activities. It will be measured daily by completion of a single question designed for the study. The question is: How important was UVR protection of your face today compared to other things you wanted/needed to do? (0=not at all - 10=very important)? Participants respond by marking a number between 0 and 10. A higher scores indicates giving protection a higher priority. Mean daily prioritisation will be recorded across each 21 day measurement period for each participant.
Mean daily self-efficacy for UVR protection in the presence of barriers | It will measured in all participants for 21 days at 3 time periods: baseline, 10 weeks and 16 weeks post baseline. The control group will complete a 21 day follow-up at 12 months (52 weeks) and 14.5 months (62 weeks) post baseline.
  This is a self reported measure of self efficacy for successfully carrying out UVR protection activities in the presence of barriers. It will be measured daily by completion of a single question designed for the study. The question is: How confident are you that you can protect your face well tomorrow, even if other things get in the way? (0=not at all - 10=very much so). Participants respond by marking a number between 0 and 10. A higher score indicates greater self- efficacy. Mean daily prioritisation will be recorded across each 21 day measurement period for each participant.
EuroQoL five dimensions scale (EQ-5D-5L) | This will be measured on single occasions: baseline, 10 weeks, 16 weeks, 36 weeks post baseline. The control group will complete follow-up at 12 months (52 weeks),14.5 months (62 weeks) and 21 months (84 weeks) post baseline.
  The EQ-5D is a standardised validated published measure of health related quality of life. It measures 5 dimensions mobility, self-care, usual activities, pain/discomfort and anxiety/depression. There are 5 responses to each domain increasing in severity (no problem to extreme problems for each domain). For each domain a higher score indicates worse health related quality of life in that domain. It also records self-rated health on a visual analogue scale (0-100), with a higher score indicating better health. A single index score can be derived from the domains giving a score between 0-1 (a higher score indicates higher health related quality of life).
4-item Self-Report Behavioural Automaticity Index (SRBAI) | This will be measured on single occasions: baseline, 10 weeks, 16 weeks, 36 weeks post baseline. The control group will complete follow-up at 12 months (52 weeks),14.5 months (62 weeks) and 21 months (84 weeks) post baseline.
  Validated published measure of automaticity of behaviour. It consists of 4 items, where the respondent rates the extent to which they agree with 4 statements related to automaticity and the behaviour (UVR protection) (e.g., UVR protection is something I do automatically (1=strongly disagree - 7=strongly agree). A composite score is the mean of the four items. A higher score indicates greater automaticity.
Short-form Warwick Edinburgh Mental Well-being scale (SWEMWBS) | This will be measured on single occasions: baseline, 10 weeks, 16 weeks, 36 weeks post baseline. The control group will complete follow-up at 12 months (52 weeks),14.5 months (62 weeks) and 21 months (84 weeks) post baseline.
  The SWEMWBS is a validated published measure of emotional wellbeing and is composed of 7 items related to a positive aspect of wellbeing (e.g., I've been feeling useful"). Respondents rate how often they have experienced each aspect over the previous 2 weeks (e.g., none of the time rarely, some of the time, often or all of the time) on a scale of 1-5. Scores are summed and then translated to a continuous metric using conversion tables (7-35). A higher score indicates higher levels of emotional wellbeing.
Photoprotection self-efficacy Questionnaire (PSEQ) | This will be measured on single occasions: baseline, 10 weeks, 16 weeks, 36 weeks post baseline. The control group will complete follow-up at 12 months (52 weeks),14.5 months (62 weeks) and 21 months (84 weeks) post baseline.
  This was developed for the study. The questionnaire assesses self-efficacy in the context of barriers using 5 items. Three items ask the respondent to rate their level of confidence that they can carry out a type of photoprotection behaviour (shifting timing or duration of outdoor activity, photoprotect using clothing, correctly apply sunscreen) on a 0-10 scale (0=Not at all - 10=very confident). Two items ask about confidence to carry out clothing protection and sunscreen application in the presence of a variety of barriers (e.g., How confident are you that you can photoprotect even if ....you are with new people?). A mean overall self-efficacy score will be calculated.
Brief Photoprotection Adherence Questionnaire (BPAQ) | This will be measured on single occasions: baseline, 10 weeks, 16 weeks, 36 weeks post baseline. The control group will complete follow-up at 12 months (52 weeks),14.5 months (62 weeks) and 21 months (84 weeks) post baseline.
  This was developed for the study as a secondary measure of photoprotection behaviour. It has 3 questions assessing frequency of protection over the previous 7 days (e.g., When you went outside, how often did you protect your face against UVR using protective clothing? 0=never - 10=all the time) and 2 questions asking about the amount of time spent out of doors during the day (never, 30 mins or less, up to 8 hours) and during periods when UVR is at its highest (11am-3pm). Items 1 to 3 are summed to give a score between 0-27, where a higher score indicates better photoprotection. Items 4 and 5, are reported individually.
Health Economic evaluation of the intervention | All participants will complete at baseline and 36 weeks post baseline. Control group will complete this at 21 months (84 weeks) post baseline.
  Financial impact of the intervention will be assessed by a questionnaire assessing health service use and the costs of XP to the participant. The questionnaire is an adapted version of the Client Service Receipt Inventory (CSRI). This retrospectively assesses use of primary and secondary healthcare services (including surgical interventions), social care, medication, tests/investigations, and aids and adaptations. Other impacts of XP measured will include time lost from work and education by patients and extra time spent caring by family members.
Mean daily dose of ultraviolet radiation (UVR) to the face using a dosimeter | It will measured in all participants for 21 days at 16 weeks post baseline
  The mean daily dose of UVR will be calculated by combining data from: (i) A UVR recorder wrist-worn device, (dosimeter) (ii) Patients' photoprotective activities self-monitored and recorded on a diary. The dosimeter provides real-time measurements of ambient UVR. It measures UVR in units of Standard Erythemal Dose (SEDs), every 5 seconds and records the mean every 5 minutes. The diary has a grid format with the day split into 15 minute segments. Participants record time spent outside rounded to the nearest 15 minutes and their photoprotection activity (e.g. hat, hoodie worn-up) during that time. During each 15 minute interval the dose of UVR to the face (in SEDs) equals the UVR exposure recorded by the dosimeter weighted by the protection associated with photoprotection behaviours recorded for that interval on the diary. Weights will be generated based on the degree of photoprotection afforded by each activity.

OTHER OUTCOMES:
Qualitative evaluation of the intervention from the perspective of the patient | They will be conducted after the 16 weeks post baseline assessement (intervention group) and post 17 months (control group)
  Semi-structured face-to-face interviews will be conducted to explore: i) the psychological mechanisms of change which explain the change in photoprotection behaviour; ii) the acceptability of the intervention from the perspective of the participant. Topics are likely to include: whether/how the intervention changed their beliefs regarding illness/treatment, confidence and motivation to photoprotect, what aspects they liked/disliked, how helpful they found the intervention, how difficult it was to make (and sustain) changes in beliefs and practices.
Self report Intervention Feedback questionnaire | It will be completed post intervention at 16 weeks follow-up (intervention group) and for the control group at 14.5 months (68 weeks)
  This is designed for this study. It has 5 items assessing overall perceptions of the programme and its components, the impact on photoprotection behaviour and whether psychosocial variables have changed as a result of the intervention. The questionnaires assesses the extent to which respondents agree with statements about the intervention (e.g., "Overall the programme was interesting/easy to understand/ helpful" 1=Strongly disagree - 5=Completely agree). A mean score of all the items will give an overall score. A higher score indicates more favourable feedback. The questionnaire will be used to inform the content of the qualitative interviews.
Profiling questionnaire | At baseline, 36 weeks post baseline. Control group will complete at 12 months (52 weeks) and 21 months (84 weeks) post baseline. Individual items will be used during qualitative interview.
  To personalise the intervention for each individual participant, a profiling questionnaire was developed for this study. The questionnaire has 21 items which assess drivers associated with suboptimal adherence to photoprotection. For example "How much do you think XP treatment at the clinic can help your skin or eye health?" (0-not at all, 10-very much). A higher score indicates greater strength of each driver. The pattern of responses will be assessed to ascertain which driver/s are important for each participant. This profile will be used to guide the content of the intervention for each participant.
Hospital Anxiety and Depression Scale (HADs) | All participants at baseline and at 12 months (52 weeks) for the control group.
  Self-reported validated published measure of Anxiety and Depression. It will be used to screen participant for clinical levels of anxiety and depression. It consists of 7 statements about anxiety and 7 about depression. Respondents are asked to indicate their agreement with the statement on a 4 point Likert scale. Scores range between 0 and 21 for each subscale. A score of 11< suggests presence of a mood disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sarkany, FRCP MD CCST, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; John Weinman, PhD, FbPsS, Principal Investigator — King's College London
Locations (1):
- Guy's St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make participant data available to other researchers.

REFERENCES:
- [Background] Walburn J, Sarkany R, Norton S, Foster L, Morgan M, Sainsbury K, Araujo-Soares V, Anderson R, Garrood I, Heydenreich J, Sniehotta FF, Vieira R, Wulf HC, Weinman J. An investigation of the predictors of photoprotection and UVR dose to the face in patients with XP: a protocol using observational mixed methods. BMJ Open. 2017 Aug 21;7(8):e018364. doi: 10.1136/bmjopen-2017-018364. PMID 28827277
- [Derived] Walburn J, Norton S, Sarkany R, Sainsbury K, Araujo-Soares V, Morgan M, Canfield M, Foster L, Heydenreich J, McCrone P, Mander A, Sniehotta FF, Wulf HC, Weinman J. Evaluation of a personalised adherence intervention to improve photoprotection in adults with Xeroderma Pigmentosum (XP): protocol for the trial of XPAND. BMJ Open. 2019 Jul 17;9(7):e028577. doi: 10.1136/bmjopen-2018-028577. PMID 31320353